CLINICAL TRIAL: NCT02185118
Title: In-vitro Experimental Study About Effects of Subanesthetic Isoflurane/Sevoflurane in 60% Oxygen on Clinical In-vitro Sepsis
Brief Title: Effects of Subanesthetic Isoflurane/Sevoflurane in 60% Oxygen on Clinical In-vitro Experimental Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Lichao Hou, M.D., Ph.D, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSFC-81171839; Chinese NSFC (Other Grant/Funding Number: 30672041, 81171839 to Lichao Hou)
Record Dates: First submitted 2014-06-20; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Oxygen; Sevoflurane; Isoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oxygen plus isoflurane/sevoflurane (Experimental): All human peripheral blood mononuclear cells (PBMCs) were from patients with non sepsis/non SIRS/non infection.
  The above cells were treated with oxygen or oxygen plus isoflurane/sevoflurane after stimulation of lipopolysaccharide/plasma from septic patients.
  Interventions: Drug: oxygen; Drug: Sevoflurane; Drug: Isoflurane

INTERVENTIONS:
Drug: oxygen — 1. Clinical in-vitro sepsis was induced in peripheral blood monocytes of non-septic patients by lipopolysaccharide or plasma from septic patients.
  2. Treatment of 100% oxygen or subanesthetic sevoflurane in 60% oxygen or subanesthetic isoflurane in 60% oxygen was performed on human peripheral blood mononuclear cells (PBMCs) stimulated by lipopolysaccharide or plasma from septic patients.
  Other Names: 100% oxygen
Drug: Sevoflurane — 1. Clinical in-vitro sepsis was induced in peripheral blood monocytes of non-septic patients by lipopolysaccharide or plasma from septic patients.
  2. Treatment of 100% oxygen or subanesthetic sevoflurane in 60% oxygen was performed on human peripheral blood mononuclear cells (PBMCs) stimulated by lipopolysaccharide or plasma from septic patients.
  Other Names: subanesthetic sevoflurane in 60% oxygen
Drug: Isoflurane — 1. Clinical in-vitro sepsis was induced in peripheral blood monocytes of non-septic patients by lipopolysaccharide or plasma from septic patients.
  2. Treatment of 100% oxygen or subanesthetic isoflurane in 60% oxygen was performed on human peripheral blood mononuclear cells (PBMCs) stimulated by lipopolysaccharide or plasma from septic patients.
  Other Names: subanesthetic isoflurane in 60% oxygen

SUMMARY:
Sepsis is a major cause of death in intensive care units. Despite the investigators improved understanding, which has reduced the risk of dying with sepsis, the number of people who die each year continues to increase due to an overall increase in the number of cases.In our previous study, the investigators have showed that 100% oxygen or 0.5 minimum alveolar concentration (MAC) isoflurane/sevoflurane in 60% oxygen protect mouse macrophage cell line against in-vitro sepsis induced by lipopolysaccharide (LPS).

In this study, the investigator hypothesized that treatment of 100% oxygen or 0.5 MAC isoflurane/sevoflurane in 60% oxygen protected against clinical in-vitro models of sepsis induced by LPS or plasma from septic patients.

DETAILED DESCRIPTION:
100% oxygen or 0.5 MAC isoflurane/sevoflurane in 60% oxygen would inhibit increases of tumor necrosis factor (TNF)-alpha, interleukin-1beta, interleukin-6 in the cell culture supernatant after stimulation of LPS or plasma from septic patients, and also inhibit the nuclear location of nuclear factor-kappa B p65 subunit.

ELIGIBILITY:
Inclusion Criteria:

* Human PBMCs were only isolated from the adult patients without sepsis/SIRS/infectious diseases.
* The plasma for induction of clinical in-vitro sepsis, was only isolated from adult patients with sepsis.

Exclusion Criteria:

* Patients who had been selected for other clinical trials in the 3 months before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Subcellular location of Nuclear Factor-KAPPA B p65 subunit | within 10 hours after the intervention

SECONDARY OUTCOMES:
tumor necrosis factor-alpha | within 10 hours after the intervention
interleukin- 1 beta | within 10 hours after the intervention
interleukin 6 | within 10 hours after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lichao Hou, M.D., Ph.D., Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Department of Anesthesiology, Xijing Hospital, Fourth Military Medical University,, Xi'an, Shaanxi, China